CLINICAL TRIAL: NCT03769220
Title: Protocol for the Method Study: Evaluation of the Measurement Properties of an Instrumented and Repeated Timed Up and Go (5iTUG)
Brief Title: Evaluation of the Measurement Properties of a 5 Time Repeated Instrumented Timed Up and Go (5iTUG)
Acronym: 5iTUG
Status: Completed | Type: Observational
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Corinna Nerz, Research associate/PhD Candidate, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Other Study IDs: 850/2018BO1
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Measurement Properties of 5iTUG; Physical Disability; Balance; Cognitive Impairment; Leg Strength; Gait Disorder, Sensorimotor; Activity of Daily Living
Keywords: Time up and Go Test
MeSH Terms: conditions — Cognitive Dysfunction; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- inpatient rehabilitation ward: The first 20 participants will be recruited from the inpatient rehabilitation ward at Robert-Bosch-Hospital (RBK). The treating medical doctor will inform potentially eligible participants about the possibility of being involved in this study. Should participants confirm their interest a research assistant will complete a detailed information session and obtain written informed consent prior enrolment.
  Participants in the study don't receive any interventions, just a baseline measurement (only health outcomes are assessed).
- outpatient rehabilitation clinic: Further 20 participants will be recruited through the outpatient rehabilitation clinic at Robert-Bosch-Hospital (RBK). The treating doctor will again inform the potential participant about the study and invite them to participate. A research assistant will complete a detailed information session and written informed consent will be obtained prior enrolment.
  Participants in the study don't receive any interventions, just a baseline measurement (only health outcomes are assessed).
- community dwelling older adults: Lastly 20 community dwelling older adults will be invited to participate. Recruitment will occur through advertisement at a locally run seniors fitness group, conducted every Thursday at RBK. Older adults who are interested in being involved will be invited to receive additional information about the study and the involved procedures before providing written informed consent and being enrolled.
  Participants in the study don't receive any interventions, just a baseline measurement (only health outcomes are assessed).

SUMMARY:
In order to tailor interventions, objective assessments of physical function is needed. A limitation of several of today's clinical assessments is that they require too much time and/or space. The Timed Up and Go (TUG) is a commonly used clinical test of physical function in older populations. The TUG is particularly useful due to its short administration time and the little space that is required. The TUG is however of limited value when used in higher-functioning older adults due to ceiling effects. Instrumented versions of TUG (iTUG) computes several outcome measures in addition to the traditional outcome measure which is the total duration. The aim of this study is to evaluate the construct- and discriminative validity of outcomes derived from sensor signals recorded with a smartphone during a five times repeated iTUG (5iTUG).

DETAILED DESCRIPTION:
At "Robert-Bosch-Krankenhaus" (RBK) in Stuttgart the investigators aim to recruit a sample consisting of 60 geriatric participants. The sample will recruited from a mix of health care settings in order to allow for cohort specific analysis.

The first 20 participants will be recruited from the inpatient rehabilitation ward at RBK. The treating medical doctor and Prof Dr Clemens Becker will inform potentially eligible participants about the possibility of being involved in this study. Should participants confirm their interest a research assistant will complete a detailed information session and obtain written informed consent prior enrolment.

Further 20 participants will be recruited through the outpatient rehabilitation clinic at RBK. The treating doctor will again inform the potential participant about the study and invite them to 6 participate. A research assistant will complete a detailed information session and written informed consent will be obtained prior enrolment.

Lastly 20 community dwelling older adults will be invited to participate. Recruitment will occur through advertisement at a locally run seniors fitness group, conducted every Thursday at RBK. Older adults who are interested in being involved will be invited to receive additional information about the study and the involved procedures before providing written informed consent and being enrolled.

All participation is entirely voluntary. Participants are free to withdraw at any time without stating a reason. Withdrawal or non-participation will not impact the care and services they are receiving or will receive from RBK now or in the future.

The following inclusion criteria will be used: community-dwelling, aged between 60 and 80 years and are able to walk 30m independently. Participants will be excluded if they report any severe cardiovascular, pulmonary, neurological, or mental diseases.

In Trondheim researchers will recruit and include 20 healthy seniors, men and women, from senior exercise groups in local fitness centres and the municipality of Trondheim. They will approach leaders or instructors of the exercise groups and ask them to contact the participants in their exercise groups to ask whether they want to take part in this study. Those who are willing will be contacted by a research coordinator. Written informed consent will be obtained prior enrolment.

Participants will be randomized to start with either the five times repeated instrumented Time up an Go Test (5iTUG) or clinical tests. The clinical tests include seven tests: the Community Balance and Mobility Scale (CBMS) (only the group of healthy participants), 8-level Balance Scale, 30s Chair stand (CS), Five times sit-to-stand (STS), Short Physical Performance Battery (SPPB), fast and habitual gait speed over 7 meters. Participants will complete the clinical tests according to the current standard clinical procedures. For the 5iTUG, participants will be instructed to do the Time up and Go Test (TUG) five times with 30 seconds rest between each repetition. The assessor will tell the participant when they should start walking. Participants will wear a smartphone attached with a belt to their lower back during the entire test sequence, both during the clinical tests and the 5iTUG. The assessor will demonstrate each test before the participants start. Participants can take breaks between tests or trials if needed. The assessor is experienced with testing of physical function in older adults, and will stand close to participants during all tasks especially where balance is challenged. At the end of the test-session, the assessor will administer one questionnaire about activities of daily living (ADL) function (the Late Life Function and Disability (LLFDI) questionnaire) and cognitive impairment based on screening via the Montreal Cognitive Assessment (MoCA).

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling
* aged between 60 and 80 years
* are able to walk 30m independently

Exclusion Criteria:

* any severe cardiovascular, pulmonary, neurological, or mental diseases.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first 20 participants will be recruited from the inpatient rehabilitation ward at Robert-Bosch-Hospital.
  Further 20 participants will be recruited through the outpatient rehabilitation clinic at Robert-Bosch-Hospital.
  Lastly 20 community dwelling older adults will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
five time repeated instrumented time up and Go Test (5iTUG) | Baseline
  Discriminative ability of the 5iTUG compared to other clinical measurements (include acceleration, velocity, duration of movements, number of steps, and step variability, from the different sub-phases of the TUG test, such as sit-to-walk, walk, first/last turn, and walk-to-sit). By performing five repetitions of an instrumented TUG (5iTUG), it is possible to get features that are more sensitive from the instrument, in addition to in total five repetitions of sit-to-stand, turning, and turn-to-sit movements, along with a total of 30 meters of walking. The 5iTUG quantifies the movement characteristics from tasks that resembles those carried out in other independent clinical measurements and test batteries, such as the Five times sit-to-stand, gait assessments, and 30s chair stand. Variability repetitions within the trials will be analysed using a repeated measures analysis.

SECONDARY OUTCOMES:
five time Sit to Stand (5xSTS) | Baseline
  needed time for 5 time repeated sit to stand
30 seconds Chair Stand (30s CS) | Baseline
  30 seconds chair stand number of repetitions
Gait speed | Baseline
  Gait speed measurement over 7 meters (habitual and fast gait speed), stopped with stopwatch
Community Balance and Mobility Scale (CBMS) | Baseline
  Community Balance and Mobility Scale, Score range from 0-96 points (with 96 is the best performance), duration: 35 minutes
8-level balance score | Baseline
  8-level balance score, each balance position held for 15 seconds, test stopped when position can not be completed, scored out of 8, higher points indicate better performance
Short Physical Performance Battery (SPPB) | Baseline
  Short Physical Performance Battery total and sub-scores, 3 balance tests each balance position held for 10 seconds, test stopped when position can not be completed, habitual gait speed over 4m, 5 time sit to stand, higher points indicate better performance, score range 0-12, duration: 8 minutes
Late Life Function and Disability questionnaire for Function (LLFDI) | Baseline
  Late Life Function and Disability (LLFDI) questionnaire, subjective measurement of functional ability and disability, scale range 0-100 points, higher points indicate better performance

CONTACTS AND LOCATIONS:
Locations (1):
- Robert-Bosch-Hospital, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Studenski S, Perera S, Wallace D, Chandler JM, Duncan PW, Rooney E, Fox M, Guralnik JM. Physical performance measures in the clinical setting. J Am Geriatr Soc. 2003 Mar;51(3):314-22. doi: 10.1046/j.1532-5415.2003.51104.x. PMID 12588574
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Schoene D, Wu SM, Mikolaizak AS, Menant JC, Smith ST, Delbaere K, Lord SR. Discriminative ability and predictive validity of the timed up and go test in identifying older people who fall: systematic review and meta-analysis. J Am Geriatr Soc. 2013 Feb;61(2):202-8. doi: 10.1111/jgs.12106. Epub 2013 Jan 25. PMID 23350947
- [Background] Mellone S, Tacconi C, Chiari L. Validity of a Smartphone-based instrumented Timed Up and Go. Gait Posture. 2012 May;36(1):163-5. doi: 10.1016/j.gaitpost.2012.02.006. Epub 2012 Mar 14. PMID 22421189